CLINICAL TRIAL: NCT02209675
Title: Role of Tissue C4d in Differentiation Between Acut e Rejection and HCV Recurrence After Liver Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Iman Fawzy Montasser, Lecturer of tropical medicine , Ain Shams university, Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: tissue C4d
Record Dates: First submitted 2014-07-31; First posted 2014-08-06 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Liver Disease
Keywords: hepatitis C recurrence; Rejection; Liver Transplantation; Liver biopsy
MeSH Terms: conditions — Liver Diseases; Rejection, Psychology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- patients with elevated liver enzymes (Other): Patients with elevated liver enzymes and/or hyperbilirubinemia post transplantation for hepatitis C virus related disease will have liver biopsy
  Interventions: Other: liver biopsy

INTERVENTIONS:
Other: liver biopsy — C4d assessment by immunohistchemistry in liver biopsy

SUMMARY:
Assessment of the role of tissue C4d complement fragments in liver biopsy as a new marker for differentiating between acute rejection and Hepatitis C (HCV) recurrence in recipients post living donor liver transplantation (LDLT) .As each condition require different treatment

DETAILED DESCRIPTION:
Role of tissue c4d assessment by immunohistchemistry in liver biopsy in differentiation between recurrent hepatitis c and rejection after liver transplantation.pathological examination may be sometimes confusing between the rejection and recurrent hepatitis C

ELIGIBILITY:
Inclusion Criteria:

* Patients transplanted for HCV related disease that are presented with elevated liver enzyme and/or hyperbilirubinemia and normal Abdominal Doppler ultrasound and Magnetic resonance cholangiography (MRCP).

Exclusion Criteria:

* Evidence of other causes of elevated liver enzyme and/or hyperbilirubinemia as abnormal Abdominal Doppler ultrasound and/or Magnetic resonance cholangiography MRCP findings.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-12; Primary Completion 2014-06 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Number of participants who developed Acute cellular rejection after transplantation | 2 years
  Assessment of the role of tissue C4d complement fragments in liver biopsy as a new marker for differentiating between acute rejection and hepatitis C recurrence in recipients post living donor liver transplantation (LDLT) .Each condition require different therapeutic management and the differentiation between them by ordinary methods is confusing due to overlapping pathological features between the rejection and recurrent hepatitis C desease

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams center for organ transplant (ASCOT), Cairo, Egypt